CLINICAL TRIAL: NCT03856073
Title: The Training and Evaluate Effect of Simulation on Clinical Airway Management for Novices During Perioperative Period
Brief Title: The Training and Evaluate Effect on Clinical Airway Management for Novices.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Chunhua Yu, Chief Physician, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: zs1809（novice）
Record Dates: First submitted 2019-02-14; First posted 2019-02-27 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Airway Management; Education; Bronchoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Novice (Experimental): Anesthesiologists without experiment of manufacturing bronchoscopy.
  Interventions: Behavioral: Novice

INTERVENTIONS:
Behavioral: Novice — Using the simulate device, the novices in bronchoscopy are going to trained and evaluated the ability of driving bronchoscopy in simulate device and clinical practice.

SUMMARY:
In this self-control experiment, anesthesiologists without experiment of bronchoscopy working in anesthesiology department in Peking Union Medical College Hospital will receive a training and evaluation procedure in simulation and clinical practice about clinical airway management. The objects was (1) to investigate the improvements of manufacturing bronchoscopy in simulation and clinical practice before and after training on simulation, (2) to record the study curve and efforts trainees needed to achieve proficiency and self-confidence on simulation, (3) to record the curve of manufacturing from skilled to unskilled, (4)to evaluate if status manufacturing on simulations could reflect the ones in clinical practice.

DETAILED DESCRIPTION:
A modified global rating scale from 1 (unskilled) to 5 (expert) with a score of 3 linked to proficiency, and 5-points Likert from 1 (felt extremely unsure) to 5 (felt extremely confidence) with a score of 4 linked to confidence were used to evaluate during the procedure of training and evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. An anesthesiologist who is working on anesthesia airway management;
2. During the research period, he/she worked in the anesthesiology department of Peking Union Medical College Hospital;
3. Have no experience of manufacturing bronchoscopy.

Exclusion Criteria:

1. Cannot complete pre-training assessment; or get more than 3 of modified global rating scale score.
2. Cannot complete the training course;
3. Cannot complete the post-training evaluation;
4. Clinical airway managers were not performed during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-03-06 (Estimated); Primary Completion 2019-05-31 (Estimated); Study Completion 2020-01-02 (Estimated)

PRIMARY OUTCOMES:
Change of Time needed. | Changes from baseline after finishing simulate training, an average of 1 month.
  Change of time needed to navigate using bronchoscopy.
Change of modified global rating scores (GRS). | Changes from baseline after finishing simulate training, an average of 1 month.
  Change of modified global rating scores (GRS) rating manufacturing skills using bronchoscopy. Total score ranges from 4 to 20 scores at 1-score intervals, higher score matches better skill. Total score is the submission of four subscales, which evaluating central view, mucosal contact, progress and orientation using bronchoscopy, ranges from 1 to 5 scores at 1-score interval, higher scores represent better outcome.
Change of Likert score. | Changes from baseline after finishing simulate training, an average of 1 month.
  Change of Likert score evaluating self-confidence using bronchoscopy. Likert score ranges from 1 to 5 scores at 1-score intervals, higher score with more self-confidence.

SECONDARY OUTCOMES:
Inconsistency of evaluation of time needed between simulate and clinical practice. | 1 day, 2 days, and every continuous 7 days until 1 month after training.
  Inconsistency of time needed to navigate using bronchoscopy.
Inconsistency of evaluation of modified global rating scores between simulate and clinical practice. | 1 day, 2 days, and every continuous 7 days until 1 month after training.
  Inconsistency of modified global rating scores (GRS) rating manufacturing skills, using bronchoscopy. Total score ranges from 4 to 20 scores at 1-score intervals, higher score matches better skill. Total score is the submission of four subscales, which evaluating central view, mucosal contact, progress and orientation using bronchoscopy, ranges from 1 to 5 scores at 1-score interval, higher scores represent better outcome.
Inconsistency of evaluation of Likert socre between simulate and clinical practice. | 1 day, 2 days, and every continuous 7 days until 1 month after training.
  Inconsistency of Likert score evaluating self-confidence using bronchoscopy. Likert score ranges from 1 to 5 scores at 1-score intervals, higher score with more self-confidence.

OTHER OUTCOMES:
Efforts needed on simulate. | An average of 6 hours, since begin of simulate training.
  Hours needed to achieve well-trained.

CONTACTS AND LOCATIONS:
Overall Officials: Chunhua Yu, Study Chair — Peking Union Medical College Hospital